CLINICAL TRIAL: NCT05188833
Title: Electrophysiological Results of the Efficacy of Deep Transcranial Magnetic Stimulation on Mood State and Quality of Life in Obsessive Compulsive Disorder Patients
Brief Title: EEG Results of Deep TMS in Patients With OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EEG.DeepTMS.OCD
Record Dates: First submitted 2021-12-26; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-10

CONDITIONS: Obsessive-Compulsive Disorder; EEG With Periodic Abnormalities
Keywords: Obsessive compulsive disorder; Deep Transcranial Magnetic Stimulation; Mood; Quality of Life; EEG
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Deep Transcranial Magnetic Stimulation (Active Comparator): The treatment will be carried out for 6 weeks, 5 days a week, in total 30 sessions; 20 hz using Brainsway H-7 helmet. It will be applied to the mPFC and ACC simultaneously with a total of 2000 beats at a frequency of 50 beats in each string.
  Interventions: Device: Deep Transcranial Magnetic Stimulation
- Deep Transcranial Magnetic Stimulation and Paroxetine (Experimental): The treatment will be carried out for 6 weeks, 5 days a week, in total 30 sessions; 20 hz using Brainsway H-7 helmet. It will be applied to the mPFC and ACC simultaneously with a total of 2000 beats at a frequency of 50 beats in each string. In addtion to DTMMS, paroxetine will applied.
  Interventions: Device: Deep Transcranial Magnetic Stimulation; Drug: Paroxetine
- Paroxetine (Active Comparator): Paroxetine is a type of antidepressant known as an SSRI (selective serotonin reuptake inhibitor). It's often used to treat depression in OCD.
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation — Deep TMS, unlike traditional TMS, is a treatment method that provides stimulation of lower parts of the brain and larger brain volume, in addition to drug treatment and psychotherapy approaches, in addition to localized brain regions magnetic stimulation is a treatment method where disease symptoms are addressed.
  Arms: Deep Transcranial Magnetic Stimulation; Deep Transcranial Magnetic Stimulation and Paroxetine
Drug: Paroxetine — Paroxetine is a type of antidepressant known as an SSRI (selective serotonin reuptake inhibitor). It's often used to treat depression.
  Arms: Deep Transcranial Magnetic Stimulation and Paroxetine; Paroxetine

SUMMARY:
Obsessive Compulsive Disorder (OCD) is a psychiatric disorder in which involuntary thoughts and irresistible behaviors are seen and its prevalence affects 2%-3% of the general population. Deep TMS is a treatment method that provides stimulation of lower parts of the brain and larger brain volume, and in addition to drug treatment and psychotherapy approaches, magnetic stimulation of localized brain regions and disease symptoms are addressed. The presence of the medial prefrontal cortex and anterior cingulate cortex in the dysfunction on the specified cycle seen in OCD patients indicates that the stimulation of these regions is necessary for a meaningful result in the treatment of deep TMS; studies show that the effect of the deep TMS method emerges as a result of the stimulation of these regions. 30 patients with OCD will included into the study and dividen into 3 groups (DTMS (n=10), DTMS + Paroxetine (n=10), Control(n=10)). Patients will evaluated in terms of depression, quality of life, and EEG before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Obsessive Compulsive Disorder within the framework of DSM-5 criteria

Exclusion Criteria:

* Not volunteering to comply with the research program
* Presence of a metal piece on the head
* Having a pacemaker inserted
* Having had a previous epileptic seizure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography | 6 weeks after baseline
  It is an electrophysiological neuroimaging method frequently used in neuroscience and clinic, in which the activity between neural circuits can be measured and observed non-invasively in the form of electrical waves.

SECONDARY OUTCOMES:
Beck Depression Scale | 6 weeks after baseline
  It is the scale used for evaluated the level of depression. Higher score means worse result.
World Health Organization Quality of Life Scale Short Form | 6 weeks after baseline
  It is the scale used for evaluated the level of quality of life. It contains a total of 26 questions. Higher score means better result.

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, PhD, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)